CLINICAL TRIAL: NCT06361875
Title: A Phase I/II Study to Investigate the Safety and Immunogenicity of Quadrivalent Influenza mRNA Vaccines MRT5421, MRT5424, and MRT5429 in Healthy Participants Aged 18 Years and Above
Brief Title: A Study to Investigate the Safety and Immunogenicity of the Quadrivalent Influenza mRNA Vaccines in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00045; U1111-1295-2852 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-04-04; First posted 2024-04-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Parallel with dose escalation for sentinel cohort
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Modified double-blind (Participants; Sites except for those preparing/administering study intervention; Sponsor's except Sponsor unblinded internal safety review committee)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Quadrivalent Influenza mRNA Vaccine MRT5421 Dose 1 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5421
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5421
- Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 1 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5429
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5429
- Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 2 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5429
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5429
- Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 3 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5429
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5429
- Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 4 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5429
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5429
- Quadrivalent Influenza mRNA Vaccine MRT5424 Dose 1 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5424
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5424
- Quadrivalent Influenza mRNA Vaccine MRT5424 Dose 2 (Experimental): participants will receive a single dose of QIV mRNA vaccine MRT5424
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5424
- Quadrivalent Influenza SD Vaccine (Active Comparator): participants will receive a single dose of QIV-SD vaccine
  Interventions: Biological: Quadrivalent Influenza Standard Dose Vaccine
- Quadrivalent Influenza HD Vaccine (Active Comparator): participants will receive a single dose of QIV -HD vaccine (for adults ≥ 65 years of age only)
  Interventions: Biological: Quadrivalent Influenza High-Dose Vaccine
- Quadrivalent Influenza RIV4 Vaccine (Active Comparator): participants will receive a single dose of RIV4 vaccine
  Interventions: Biological: Quadrivalent Recombinant Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza mRNA Vaccine MRT5421 — Pharmaceutical form:solution in a vial-Route of administration:Intramuscular injection
  Arms: Quadrivalent Influenza mRNA Vaccine MRT5421 Dose 1
Biological: Quadrivalent Influenza mRNA Vaccine MRT5424 — Pharmaceutical form:solution in a vial-Route of administration:Intramuscular injection
  Arms: Quadrivalent Influenza mRNA Vaccine MRT5424 Dose 1; Quadrivalent Influenza mRNA Vaccine MRT5424 Dose 2
Biological: Quadrivalent Influenza mRNA Vaccine MRT5429 — Pharmaceutical form:solution in a vial-Route of administration:Intramuscular Injection
  Arms: Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 1; Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 2; Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 3; Quadrivalent Influenza mRNA Vaccine MRT5429 Dose 4
Biological: Quadrivalent Influenza Standard Dose Vaccine — Pharmaceutical form: suspension for injection in prefilled syringe -Route of administration:Intramuscular injection
  Other Names: Fluzone Qudrivalent®
  Arms: Quadrivalent Influenza SD Vaccine
Biological: Quadrivalent Influenza High-Dose Vaccine — Pharmaceutical form:suspension for injection in pre filled syringe -Route of administration:Intramuscular injection
  Other Names: Fluzone High-Dose Quadrivalent®
  Arms: Quadrivalent Influenza HD Vaccine
Biological: Quadrivalent Recombinant Influenza Vaccine — Pharmaceutical form:suspension for injection in pre filled syringe-Route of administration:Intramuscular injection
  Other Names: Flublok Quadrivalent®
  Arms: Quadrivalent Influenza RIV4 Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single intramuscular (IM) injection of different formulations of Quadrivalent Influenza Vaccine (QIV) messenger ribonucleic acid (mRNA) (MRT5421, MRT5424, and MRT5429) compared to an active control (QIV- standard dose (SD), QIV- high dose (HD) [adults ≥ 65 years of age only], or quadrivalent recombinant influenza vaccine (RIV4)) in adults 18 years of age and older.

DETAILED DESCRIPTION:
Study duration per participant is approximately 12 months.

* Treatment duration: 1 injection of one of the 7 QIV mRNA or one of the controls
* Dose escalation with sequential enrollment

ELIGIBILITY:
Inclusion Criteria: - Aged from 18 years on the day of inclusion or aged from 21 years on the days of inclusion, depending on the countries.

* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR
  * Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.
* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before the 1st dose of study intervention Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA vaccine
* Previous history of myocarditis, pericarditis, and / or myopericarditis
* Known history of previous episodes of Gillian-Barre Syndrome (GBS), neuritis (including Bell's palsy), convulsions, encephalitis, transverse myelitis, and vasculitis
* Participants with an ECG that is consistent with possible myocarditis or pericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Self-reported thrombocytopenia, contraindicating Intramuscular vaccination based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating Intramuscular vaccination based on Investigator's judgment
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness / infection (according to Investigator's judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Participant who had acute infection symptoms or a positive SARS-CoV-2 RT-PCR or antigen test in the past 10 days prior to the 1st visit (V01)
* Receipt of any vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine in the 4 weeks following study intervention administration
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Previous vaccination against influenza in the previous 6 months with an investigational or marketed vaccine
* Receipt of any mRNA vaccine/product in the 2 months preceding study intervention administration NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate unsolicited systemic adverse events (AEs) | Within 30 minutes after injection
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions | Up to 7 days after injection
  Adverse reactions pre-listed in the protocol and case report form (CRF) Injection site reactions: Injection site pain, Injection site erythema, and Injection site swelling
Number of participants with solicited systemic reactions | Up to 7 days after injection
  Adverse reactions pre-listed in the protocol and case report form (CRF) Systemic reactions: fever, headache, fatigue, myalgia, arthralgia, chills
Number of participants with unsolicited AEs | Up to 28 days after injection
  AEs that do not fulfill the conditions of solicited reactions
Number of participants with medically attended adverse events (MAAEs) | Up to 180 days after injection
  MAAEs reported up to 180 days after injection
Number of participants with serious adverse events (SAEs) | Throughout the study (approximately 12 months)
  SAEs reported throughout the study
AESIs reported throughout the study | AESIs reported throughout the study (approximatley 12 months)
  AESIs reported throughout the study (approximately 12 months)
Number of participants with adverse events of special interests (AESIs) | Throughout the study (approximately 12 months)
  AESIs reported throughout the study
Number of participants with out-of-range biological test results | Up to 8 days after injection
  Out-of-range biological test results (including shift from baseline values)
Geometric Mean Titer (GMT) | At Day 1 and Day 29
  Hemagglutinin inhibition (HAI) antibody (Ab) titers at D01 and D29
Geometric Mean of individual Titer Ratio (GMTR) | At Day 1 and Day 29
  Individual HAI Ab titer ratio D29/D01
Seroconversion | At Day 1 and Day 29
  Number of participants with HAI Ab titer < 10 [1/dil] at Day 1 and post-vaccination titer ≥ 40 [1/dil] at Day 29, or titer ≥ 10 [1/dil] at Day 1 and a ≥ 4-fold-rise in titer [1/dil] at Day 29
HAI Ab titer ≥ 40 (1/dil) | Day 29
  HAI Ab titer ≥ 40 (1/dil) at D29

SECONDARY OUTCOMES:
Neutralizing Ab titers at D01 and D29 | At Day 1 and Day 29
  Neutralizing Ab titers at D01 and D29
Individual neutralizing antibodies titer ratio | At Day 1 and Day 29
  Individual neutralizing antibodies titer ratio D29/D01
2-fold and 4-fold increase in neutralizing titers | Day 1 through Day 29
  2-fold and 4-fold increase in neutralizing titers

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Long Beach Clinical Trials Site Number : 8400013, Long Beach, California
  - California Research Foundation Site Number : 8400038, San Diego, California
  - Accel Clinical Research-Deland Clinical Research Unit- Site Number : 8400001, DeLand, Florida
  - SIMEDHealth, LLC- Site Number : 8400011, Gainesville, Florida
  - Indago Research and Health Center- Site Number : 8400032, Hialeah, Florida
  - Cenexel Research Centers of America- Site Number : 8400037, Hollywood, Florida
  - Suncoast Research Group, LLC- Site Number : 8400015, Miami, Florida
  - Brengle Family Medicine Site Number : 8400045, Indianapolis, Indiana
  - AMR Lexington- Site Number : 8400042, Lexington, Kentucky
  - Velocity Clinical Research- New Orleans Site Number : 8400053, New Orleans, Louisiana
  - The Alliance for Multispecialty Research - KCM, LLC- Site Number : 8400034, Kansas City, Missouri
  - Velocity Clinical Research Norfolk- Site Number : 8400046, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha- Site Number : 8400008, Omaha, Nebraska
  - Rochester Clinical Research. Inc.- Site Number : 8400005, Rochester, New York
  - Coastal Carolina Research Center- Site Number : 8400014, North Charleston, South Carolina
  - AMR Knoxville- Site Number : 8400043, Knoxville, Tennessee
  - Clinical Trials of Texas, Inc. - PPDS- Site Number : 8400029, San Antonio, Texas
  - Cenexel JBR- Site Number : 8400051, Salt Lake City, Utah
- Investigational Site Number : 3400001, San Pedro Sula, Honduras
- Investigational Site Number : 6300002, Barrio Sabana, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org